CLINICAL TRIAL: NCT03396497
Title: A Multicenter, Open-Label Study of LYC-55716 in Combination With Pembrolizumab in Adult Subjects With Metastatic Non-Small Cell Lung Cancer
Brief Title: Study of LYC-55716 With Pembrolizumab in Adult Subjects With Non-Small Cell Lung Cancer
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Lycera Corp. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LYC-55716-1002
Record Dates: First submitted 2018-01-03; First posted 2018-01-11 (Actual); Last update posted 2019-09-25 (Actual); Status verified 2019-09

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — cintirorgon; pembrolizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- LYC-55716 + pembrolizumab (Experimental): Subjects will receive combination treatment until disease progression or unacceptable toxicity, or up to a maximum of 24 months.
  Interventions: Drug: LYC-55716; Drug: Pembrolizumab

INTERVENTIONS:
Drug: LYC-55716 — Continuous twice daily administration of LYC-55716 in 28 day treatment cycles.
Drug: Pembrolizumab — Pembrolizumab administered every 3 weeks as prescribed as standard of care by the investigator in accordance with the package insert.

SUMMARY:
This is a Phase 1B study designed to assess the safety and tolerability of LYC-55716 given in combination with pembrolizumab to subjects with metastatic NSCLC, and to assess the combination for biologic and clinical activity in NSCLC.

DETAILED DESCRIPTION:
Approximately 18 subjects across 5 US sites will be enrolled in the study.

Subjects will enter a screening period of up to 28 days, followed by continuous twice daily administration of LYC-55716 in 28 day treatment cycles. Subjects will also be administered pembrolizumab every 3 weeks as prescribed as standard of care by the Investigator in accordance with the package insert.

The study will begin with a run-in cohort of 3 subjects to assess the safety and tolerability of the LYC-55716/pembrolizumab combination. Subjects in the run-in cohort will be enrolled singly at intervals of not less than 7 days in order to monitor for adverse reactions to the combination. If no subjects in the run-in cohorts has a DLT, then the study may proceed to the main cohort (15 subjects).

Subjects will receive combination treatment until clinically significant disease progression or unacceptable toxicity, or up to a maximum of 24 months.

Primary Study Objectives:

Run-in Cohort

* Evaluate the safety and tolerability of the LYC-55716/pembrolizumab combination
* Determine the dose of LYC-55716 that is adequately tolerated when used in combination with pembrolizumab

Main Study Cohort

• Further evaluate the safety and tolerability of the LYC-55716/pembrolizumab combination

Secondary Study Objectives:

Main Study Cohort

* Evaluate the cellular immune response in paired tumor biopsy samples
* Evaluate effects on circulating biomarkers in the blood of LYC-55716 with pembrolizumab
* Determine the objective response rate
* Determine the duration of response
* Determine the progression-free survival (PFS) and overall survival (OS)

ELIGIBILITY:
Inclusion Criteria:

* Subject has histologic or cytologic confirmation of metastatic NSCLC. Subjects must have a TPS score available as determined by an FDA approved test. Subject has stable disease or disease progression and is being treated with pembrolizumab therapy as standard of care by the Investigator.
* Subject is male or female and at least 18 years of age.
* Subject has at least 1 measurable lesion per RECIST v1.1 criteria by computed tomography (CT) scan or magnetic resonance image (MRI).
* Subject provides consent for fresh paired tumor biopsy samples to be obtained at screening and after 4 weeks of treatment (not required for run-in cohort or expansion of run-in cohort).
* Subject has a life expectancy of at least 12 weeks
* Subject has adequate organ function as determined by the following laboratory values:

  * ANC* ≥ 1500/mm³ (≥ 1.5 x 10^9/L)
  * Platelets* ≥ 100,000/mm³ (≥ 100 x 10^9/L)
  * Lymphocytes* ≥ 500/mm³ (≥ 0.5 x 10^9/L)
  * Hemoglobin* ≥ 9.0 g/dL
  * Serum Creatinine or Creatinine Clearance** ≤ 1.5 x ULN, > 50 mL/min
  * Total Serum Bilirubin ≤ 1.5 x ULN (< 3.0 mg/dL if subject has Gilbert's syndrome)
  * Liver Transaminases (ALT/AST) ≤ 2.5 x ULN, ≤ 5.0 x ULN if liver metastases present

    * (* = without ongoing growth factor or transfusion support)
    * (** = calculated by Cockcroft and Gault's formula)
    * (ALT = alanine aminotransferase, AST = aspartate aminotransferase, ULN = upper limit of normal)

Exclusion Criteria:

* Subjects may not have genomic aberrations such as ALK, EGFR, or BRAF for which there are FDA-approved targeted therapies available. Subjects may not have ROS1 aberration in accordance with the pembrolizumab label.
* Subject has received an investigational drug in the 28 day period before the first dose of study drug (or within 5 half-lives if longer) or is currently participating in another interventional clinical trial.
* Subject has known symptomatic brain metastases or leptomeningeal involvement as assessed by CT scan or MRI. Subjects with stable asymptomatic brain metastases or leptomeningeal disease are eligible provided that they have not required new treatments for this disease in a 28 day period before the first dose of study drug, and anticonvulsants and steroids have not been administered for a period of 2 weeks prior to the first dose of study drug.
* Subject has not recovered from adverse reactions to prior cancer treatment or procedures (surgery, chemotherapy, immunotherapy, radiation therapy) to CTCAE Grade 2 or better.
* Subject has a previous (within 5 years) or current malignancy other than the target cancer with the exception of curatively treated local tumors such as carcinoma in situ of the breast or cervix, basal or squamous cell carcinoma of the skin, or prostate cancer with Gleason Grade < 6 and prostate-specific antigen within normal range.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2018-08-03 (Actual); Primary Completion 2019-10-20 (Estimated); Study Completion 2019-10-20 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability will be assessed by the number of subjects with any treatment-emergent Adverse Events | 12 weeks
  Common terminology criteria for adverse events (CTCAE) will be used for AE assessment.

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Lycera Investigational Site, Aurora, Colorado
  - Lycera Investigational Site, Ann Arbor, Michigan
  - Lycera Investigational Site, Nashville, Tennessee
  - Lycera Investigational Site, Seattle, Washington